CLINICAL TRIAL: NCT02826499
Title: Comparison of the Malposition Rates of the Vertebral Pedicle Screws Using the PediGuard Technique: PediGuard Technique Associated With Fluoroscopy and Fluoroscopy Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tamas Illes, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUB-Pediguard
Record Dates: First submitted 2016-06-24; First posted 2016-07-11 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Pedicular Screwing
Keywords: Pediguard; Pedicular screws; Fluoroscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoroscopy (Active Comparator): Vertebral instrumentation with pedicular screwing, performed under fluoroscopy.
  Interventions: Other: Fluoroscopy
- Fluoroscopy and Pediguard (Experimental): Vertebral instrumentation with pedicular screwing, performed under fluoroscopy, with the Pediguard system.
  Interventions: Device: Pediguard; Other: Fluoroscopy

INTERVENTIONS:
Device: Pediguard — It is a guide for the perforation of the pedicular channel, with a probe at its extremity. This probe allows a real time measurement of the electric conductivity of the tissues that are being crossed. The conductivity measure is translated in a sound signal. Because the cortical bone has a low conductivity, the probe will emit a low intensity sound signal. The cancellous bone has a medium conductivity. Therefore, the probe will emit a medium sound signal. However, in the event of a breach in the pedicular cortical, as blood and periost have a high conductibility, the probe will emit a intense, rapid pace, sound signal.The Pediguard technique helps thus to anticipate a cortical effraction, by detecting the proximity of the cortical wall.
  Arms: Fluoroscopy and Pediguard
Other: Fluoroscopy — The placing of pedicular screws under fluoroscopic control is the most common technique as it is both reproducible and accessible. It is a two dimensional imaging technique. The profile incidence at the level of the spine is mostly used to spot the vertebral pedicle and the direction of the screw in the sagittal plane. However, there is no real control of the direction of the pedicular screw in the horizontal or frontal plane and it is an irradiating imaging technique.

SUMMARY:
Pedicular screwing has become the gold standard for intervertebral fixation required in degenerative, scoliotic, tumoral pathologies or for fractures. Several pedicular screwing methods exist.

The free hand pedicular screwing requires a high learning curve and has, as a consequence, a high malposition rate.

The placing of pedicular screws under fluoroscopic control is the most common technique as it is both reproducible and accessible. It is a two dimensional imaging technique. The profile incidence at the level of the spine is mostly used to spot the vertebral pedicle and the direction of the screw in the sagittal plane. However, there is no real control of the direction of the pedicular screw in the horizontal or frontal plane. The screw malposition rate is less important than with the 'free hand' technique but remains none of the less significant. Furthermore, fluoroscopy is an irradiating imaging technique, both for the patient and the staff.

New revolutionary techniques as the tridimensional navigation and the per-operatory tomodensitometry appeared in the last few years. The techniques give the best results when used concommitantly. The material has the advantage of being very precise. The pedicular screw malposition rate is minimal after a three-dimensional localisation. However, those systems require qualified staff and expose the patient and the nursing team to high radiation levels. The costs are higher and the surgery duration is globally longer. It is thus difficult to implement this technique in each belgian hospital.

Finally, the Pediguard technique appeared on the market. It is a guide for the perforation of the pedicular channel, with a probe at its extremity. This probe allows a real time measurement of the electric conductivity of the tissues that are being crossed. The conductivity measure is translated in a sound signal. Because the cortical bone has a low conductivity, the probe will emit a low intensity sound signal. The cancellous bone has a medium conductivity. Therefore, the probe will emit a medium sound signal. However, in the event of a breach in the pedicular cortical, as blood and periost have a high conductibility, the probe will emit a intense, rapid pace, sound signal.The Pediguard technique helps thus to anticipate a cortical effraction, by detecting the proximity of the cortical wall. It is efficient but remains relatively expensive.

The main objective of this study is to determine the precision of the placing of pedicular screws, with and without Pediguard system, under fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* All patients needing vertebral instrumentation with pedicular screwing

Exclusion Criteria:

* Contra-indication to the placement of pedicular screws under fluoroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pedicular effraction grade | Between 24 and 48h after surgery
  Evaluation of screw malposition, performed under CT-scan and graded according to the following: 0 (no effraction), grade 1 (effraction up to 2 mm), grade 2 (effraction between 2 and 4 mm), grade 3 (effraction of more than 4 mm).
Pedicular effraction grade | 1 year after surgery
  Evaluation of screw malposition, performed under CT-scan and graded according to the following: 0 (no effraction), grade 1 (effraction up to 2 mm), grade 2 (effraction between 2 and 4 mm), grade 3 (effraction of more than 4 mm).

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline
  Clinical functional scoring, assessed before the surgical intervention.
Oswestry Disability Index (ODI) | 1 year after surgery
  Clinical functional scoring
SF-36 questionnaire | Baseline
  Quality of life evaluation, assessed before the surgical intervention.
SF-36 questionnaire | 1 year after surgery
  Quality of life evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Illes, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium